CLINICAL TRIAL: NCT06282159
Title: A Phase 2, Randomized, Blinded, Placebo-Controlled, Study to Evaluate Safety, Tolerability, Pharmacometrics, and Efficacy of DNTH103 in Adults With Generalized Myasthenia Gravis (MAGIC)
Brief Title: A Phase 2 Study to Evaluate DNTH103 in Adults With Generalized Myasthenia Gravis (MAGIC)
Acronym: MAGIC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dianthus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNTH103-MG-201; 2024-512865-15-00 (EU CTIS Number)
Record Dates: First submitted 2023-12-15; First posted 2024-02-28 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Myasthenia Gravis, Generalized
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- DNTH103 low dose Q2W (Experimental)
  Interventions: Drug: DNTH103
- DNTH103 high dose Q2W (Experimental)
  Interventions: Drug: DNTH103

INTERVENTIONS:
Drug: DNTH103 — Day 1: IV loading dose Week 1 to Week 11: DNTH103 administered SC every 2 weeks
  Other Names: Claseprubart
  Arms: DNTH103 high dose Q2W; DNTH103 low dose Q2W
Drug: Placebo — Day 1: IV infusion of placebo Week 1 to Week 11: placebo administered SC every 2 weeks
  Arms: Placebo

SUMMARY:
The purpose of this Phase 2 study is to evaluate the safety, tolerability, pharmacometrics, and efficacy of DNTH103 in participants with generalized myasthenia gravis (gMG).

DETAILED DESCRIPTION:
The study includes the following periods:

* Screening (up to 10 weeks)
* Randomized, blinded, controlled treatment (RCT) period (13 weeks)
* Open-label extension (OLE) period (optional) for eligible participants (52 weeks)
* Safety follow-up (40 weeks)

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out.
2. Adult males and females, 18 to 75 years of age (inclusive) at Screening.
3. Weight range between 40-120 kg at Screening.
4. Diagnosis of gMG by the following tests:

   Acetylcholine receptor antibody (AChR Ab) positive, and

   One of the following:

   i. History of abnormal neuromuscular transmission test; ii. History of positive anticholinesterase test; iii. Clinical response to acetylcholinesterase inhibitors.
5. Myasthenia Gravis Foundation of America (MGFA) Class II-Iva
6. Myasthenia Gravis Activities of Daily Living (MG-ADL) score of 6 or more
7. Vaccination against N. meningitidis with the quadrivalent meningococcal vaccine, and where available, meningococcal serotype B vaccine within 3 years prior to, or at the time of, initiating study drug.
8. Female participants must:

   Be of non-childbearing potential, or if of childbearing potential, must agree not to donate ova, not to attempt to become pregnant and, if engaging in sexual intercourse with a male partner, must agree to use a highly effective method of contraception.
9. Male participants must be surgically sterile for at least 90 days prior to screening or agree not to donate sperm

Exclusion Criteria:

1. History or presence of significant medical/surgical condition including any acute illness or major surgery considered to be clinically significant
2. Prior history (at any time) of N. meningitidis infection.
3. Positive test results for active human immunodeficiency virus (HIV-1 or HIV-2), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies during Screening.
4. Any thymic surgery/biopsy within 1 year of Screening.
5. Any known or untreated thymoma.
6. Any history of thymic carcinoma or thymic malignancy.
7. Concurrent or previous use of the following medication within the time periods specified below.

   1. Rituximab within 6 months (180 days) prior to randomization (Day 1);
   2. Intravenous immunoglobulin (IVIg) and plasma exchange (PLEX) within 4 weeks (28 days) prior to randomization (Day 1).
8. Participation in another clinical study of an investigational drug within 90 days or 5 half-lives of the investigational agent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (SAEs) | Baseline (Day 1) to Week 13
  Number of participants with TEAEs and treatment-emergent SAEs will be reported.

SECONDARY OUTCOMES:
Change from Baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) Scale Score | Baseline (Day 1) to Week 13
  The MG-ADL score is an 8-item patient reported outcome (PRO) instrument. The MG-ADL targets symptoms of disability across ocular, bulbar, respiratory, and axial symptoms. The item responses are scored from 0 to 3, and the total score of the MG-ADL is the sum of the 8 items and ranges from 0 to 24, with a higher score indicating more disability.
Change from Baseline in Quantitative Myasthenia Gravis (QMG) Scale Score | Baseline (Day 1) to Week 13
  The QMG is a clinician-reported assessment to evaluate muscle strength. The QMG consists of 13 items that measure endurance or fatiguability, with each item having a possible score that ranges from 0 - 3. The total possible QMG scores range from 0 - 39, with a higher score indicating greater disease burden.
Change from Baseline to Week 13 in Myasthenia Gravis Composite (MGC) Scale Score | Baseline (Day 1) to Week 13
  The MGC is a validated assessment tool for measuring clinical status of participants with MG. The range of total MGC score is 0 to 50, with higher scores indicating more severe disease. A clinically meaningful improvement is reflected by a 3-point improvement in MGC score. The MGC assesses 10 important functional areas most frequently affected by MG and the scales are weighted for clinical significance that incorporates patient-reported outcomes.
Incidence of TEAEs and Treatment-Emergent SAEs | Baseline (Day 1) up to Week 52 of the OLE
  Number of participants with TEAEs and treatment-emergent SAEs will be reported.
Serum Concentrations of DNTH103 | Baseline (Day 1) to Week 52 of the OLE
  Blood samples will be collected for measurement of serum concentrations of DNTH103 at various timepoints both pre- and post-dose.
Change from Baseline in Complement Total Blood Test (CH50) | Baseline (Day 1) to Week 52 of the OLE
  Blood samples will be collected to determine changes in CH50 at various timepoints.
Incidence and Titer of Antidrug Antibody (ADAs) Against DNTH103 | Baseline (Day 1) to Week 52 of the OLE
  Blood samples will be collected to measure ADA against DNTH103 at various timepoints.

CONTACTS AND LOCATIONS:
Locations (50):
- United States (20):
  - Clinical Study Site, Phoenix, Arizona
  - Clinical Study Site, Irvine, California
  - Clinical Study Site, Stamford, Connecticut
  - Clinical Study Site, Boca Raton, Florida
  - Clinical Study Site, Bradenton, Florida
  - Clinical Study Site, Maitland, Florida
  - Clincal Study Site, Tampa, Florida
  - Clinical Study Site, O'Fallon, Illinois
  - Clinical Study Site, Kansas City, Kansas
  - Clinical Study Site, Lexington, Kentucky
  - Clinical Study Site, Boston, Massachusetts
  - Clinical Study Site, East Lansing, Michigan
  - Clinical Study Site, Columbia, Missouri
  - Clinical Study Site, Cincinnati, Ohio
  - Clinical Study Site, Columbus, Ohio
  - Clinical Study Site, Dallas, Texas
  - Clinical Study Site #2, Houston, Texas
  - Clinical Study Site, Houston, Texas
  - Clinical Study Site, Lubbock, Texas
  - Clinical Study Site, Richmond, Virginia
- Argentina (4):
  - Clinical Study Site, San Miguel de Tucumán, Tucumán Province
  - Clinical Study Site, Buenos Aires
  - Clinical Study Site, Córdoba
  - Clinical Study Site, Rosario
- Clinical Study Site, London, Ontario, Canada
- Clinical Study Site, Ostrava, Czechia
- Clinical Study Site, Copenhagen, Denmark
- France (3):
  - Clinical Study Site, Bordeaux
  - Clinical Study Site, Nice
  - Clinical Study Site, Strasbourg
- Israel (3):
  - Clinical Study Site, Haifa
  - Clinical Study Site, Ramat Gan
  - Clinical Study Site, Safed
- Italy (4):
  - Clinical Study Site, Milan
  - Clinical Study Site, Napoli
  - Clinical Study Site, Pisa
  - Clinical Study Site, Rome
- Clinical Study Site, Amsterdam, Netherlands
- Clinical Study Site, Skopje, North Macedonia
- Clinical Study Site, Bergen, Norway
- Poland (5):
  - Clinical Study Site, Bydgoszcz
  - Clinical Study Site, Katowice
  - Clinical Study Site, Krakow
  - Clinical Study Site, Lublin
  - Clinical Study Site, Warsaw
- Serbia (4):
  - Clinical Study Site, Belgrade
  - Clinical Study Site, Kragujevac
  - Clinical Study Site, Niš
  - Clinical Study Site, Novi Sad
- Clinical Study Site, Malmo, Sweden